CLINICAL TRIAL: NCT02748343
Title: The Clinical Therapeutic Effects and Safety of Tissue-engineered Bone
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bilong11
Record Dates: First submitted 2016-03-09; First posted 2016-04-22 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-03

CONDITIONS: Bone Defect; Bone Nonunion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- allograft bone (Active Comparator): traditional allograft bone
  Interventions: Device: allograft bone
- tissue-engineered bone (Experimental): tissue-engineered bone
  Interventions: Device: tissue-engineered bone

INTERVENTIONS:
Device: allograft bone — Use of the allograft bone to treat the bone defect in patients
  Arms: allograft bone
Device: tissue-engineered bone — Use of the tissue-engineered bone to treat the bone defect in patients
  Arms: tissue-engineered bone

SUMMARY:
The purpose of this study is to compare use of a tissue-engineered bone to use of a standard allograft bone to treat bone defect in patients. The hypothesis is that use of the tissue-engineered bone is effective and safe to treat the bone defect in patients.

DETAILED DESCRIPTION:
Patients with the bone defect without infection and sever system diseases will be recruited.

The material selected as the scaffold for this study will be a porous β-tricalcium phosphate scaffold (β-TCP) scaffold and scaffold is custom-made according to the size and shape of bone defect after three-dimensional CT scan. Human BMSCs will be obtained and cultured before operation and 3.4×106 cells in 10ml serum-free medium will be seeded onto scaffold to construct the tissue engineered bone graft and co-cultured for two weeks.

The implant operation will be carried out under the general anesthesia. The tissue engineered bone graft will be implanted into the bone defect area. The bone defect area will be covered with surrounding soft tissue and muscle to close the wound. Anti-inflammatory, repercussive and analgesic drugs will be used for 1 week.

Patient will be hospitalized for 1 to 2 weeks after surgery. Blood routine examination, erythrocyte sedimentation rate, immunoglobulin, autoantibodies and clinical examination will be carried out for signs of pain, swelling, immune rejection and infection. Patient will be evaluated at 3 days，3, 6, 12, 18 and 22 months after operation by radiography; Three-dimensional CT scan will be also performed at regular intervals. The function of the body will be evaluated at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* the patients with bone defect and bone nonunion caused by tumor or trauma
* the length of bone defect in long diaphysis is more than 4cm or more than half of the shaft diameter
* the size of bone defect is more than 5cmx5cm
* the patients are unable to use autologous bone graft or other treatments
* the patients request to use the treatment of tissue-engineered bone
* Supportive family with willingness to participate in completing questionnaires

Exclusion Criteria:

* Patients with serious diseases such as hemorrhagic disorders, infection, tumor, contagion and so on.
* Patients who are pregnant
* Patients with serious abnormal cardiopulmonary function
* Patients disagree to use the tissue-engineered bone
* Patients are older than 60 years
* Patients who are regarded to be unqualified by investigator

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The scores of bone healing | within 48 weeks after surgical treatment of bone dect
  The scores of bone healing are divided into three kinds: nonhealing: 0; delayed healing: 1; normal healing: 2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
the adverse event incidence using tissue-engineered bone and allograft bone | within 24 weeks after surgical treatment of bone dect
  the adverse event incidence of tissue-engineered bone is compared with the adverse event incidence of allograft bone to verify the safety of tissue-engineered bone.

SECONDARY OUTCOMES:
The scores of blood routine test | within 48 weeks after surgical treatment of bone dect
  The scores of blood routine test after operation are divided into three kinds: severely abnormal：0；abnormal：1；normal：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of erythrocyte sedimentation rate(ESR) | within 48 weeks after surgical treatment of bone dect
  The scores of erythrocyte sedimentation rate (ESR) after operation are divided into three kinds: severely abnormal：0；abnormal：1；normal：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of C-reactive protein | within 48 weeks after surgical treatment of bone dect
  The scores of C-reaction protein after operation are divided into three kinds: severely abnormal：0；abnormal：1；normal：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of the ratio of complement C3 to complement C4 | within 48 weeks after surgical treatment of bone dect
  The scores of ratio of complement C3 to C4 after operation are divided into three kinds: severely abnormal：0；abnormal：1；normal：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of immunoglobulin assay | within 48 weeks after surgical treatment of bone dect
  The scores of immunoglobulin assay (IgG, IgA and IgM) after operation are divided into three kinds: severely abnormal：0；abnormal：1；normal：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of duration of hospital stay | within 48 weeks after surgical treatment of bone dect
  The scores of duration of hospital stay are divided into four kinds: longer than one months: 0; longer than two weeks:1; longer than one week:2; less than one week:3. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
the scores of time of weight loading after operation | within 48 weeks after surgical treatment of bone dect
  The scores of time of weight loading after operation are divided into three kinds: longer than six months: 0; longer than three months:1; less than three months:2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of tumorigenesis | within 48 weeks after surgical treatment of bone dect
  The scores of tumorigenesis after operation are divided into three kinds: severely abnormal：0；abnormal：1；normal：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of treatment course | within 48 weeks after surgical treatment of bone dect
  The scores of treatment course are divided into three kinds: long：0；general ：1；short：2. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of number of operations | within 48 weeks after surgical treatment of bone dect
  The scores of number of operations are divided into four kinds: above three times：0； three times：1；two times：2；one time：3. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of pain | within 48 weeks after surgical treatment of bone dect
  The scores of pain after operation are divided into four kinds: severe:0;moderate:1;slight:2; none:3. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.
The scores of wound healing of soft tissue | within 48 weeks after surgical treatment of bone dect
  The scores of wound healing are divided into four kinds: infection: 0; no healing: 1; delayed healing: 2; normal healing: 3. The average score of tissue-engineered bone is compared with the score of control group using allograft bone to verify the clinical efficacy of tissue-engineered bone.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Xijing Hospital, The Fourth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided